CLINICAL TRIAL: NCT03445403
Title: Offset Analgesia as a Measure of Central Sensitization in Children With Chronic Pain Disorders
Brief Title: Offset Analgesia as a Measure of Central Sensitization in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Navil Sethna, MD, Clinical Director, Mayo Family Pediatric Pain Rehabilitation Center, Professor of Anesthesiology Harvard Medical School, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: P00025596
Record Dates: First submitted 2018-02-05; First posted 2018-02-26 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Chronic Pain Syndrome; Chronic Daily Headache; Functional Abdominal Pain Syndrome; Musculoskeletal Pain Disorder; CRPS (Complex Regional Pain Syndromes)
Keywords: Offset analgesia; Quantitive sensory testing
MeSH Terms: conditions — Headache Disorders; Collagen Diseases; Complex Regional Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Response to a moderate heat pain [defined as a heat stimulus producing pain rated at 50mm on a scale of 0-100 mm] applied the the skin of the forearm using a paradigm known as offset analgesia will be compared in children with chronic pain disorders and healthy, age and sex matched controls.
Who Masked: Participant, Outcomes Assessor
Masking Description: During offset analgesia testing, participants will be exposed to 3 heat pain paradigms: a constant heat stimulus, the offset analgesia paradigm, and a control paradigm. The participants will not be aware of the direction/pattern of temperature changes or which paradigm is being applied. Participants will not be allowed to view the computer screen so that it would not influence their response. The statistician will be unaware of the participants allocation of children with chronic pain vs. control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic pain disorders (Experimental): Administration of offset analgesia and control and constant paradigms using moderate heat pain as determined by the individual subject reporting of 50 mm on a visual analog pain scale of 0-100 mm.
  Interventions: Other: Offset analgesia
- Healthy controls (Active Comparator): Administration of offset analgesia and control and constant paradigms using moderate heat pain as determined by the individual subject reporting of 50 mm on a visual analog pain scale of 0-100 mm.
  Interventions: Other: Offset analgesia

INTERVENTIONS:
Other: Offset analgesia — Exposure to a moderate heat-pain stimulus applied for 5 seconds, raised by 1 degree C for 5 seconds, reduced by 1 degree C, and held for 20 seconds using a computerized paradigm in order to evoke endogenous pain modulation.

SUMMARY:
Pediatric chronic pain disorders are common and consequential in Western societies, occurring in 25-80% of population-based samples with a median prevalence of 11-38% and significant pain-related disability in 3-5% of these children. Pediatric chronic pain disorders have a negative impact on many aspects children's lives including mobility, night sleep, school attendance, peer relationships, family functioning, and overall quality of life. Parents caring for these children risk loss of parental earnings, and these disorders place a high financial burden on healthcare. In a nationally representative sample in the United States, costs related to health care were significantly higher ($1,339 per capita) for children with chronic pain disorders compared to children with common pediatric health conditions of ADHD, asthma and obesity.

In children with clinical chronic pain conditions, such as daily headaches or fibromyalgia, chronic pain is presumably a persistent state of an overly excitable nervous system. This phenomenon known as central sensitization is characterized by excessive pain sensitivity that occurs in response to non-painful stimuli, such as light touch or contact with clothing, and slightly painful stimuli, such as a light pinprick. This hypersensitivity results from peculiar changes in the working of the central nervous system, including the spinal cord and brain, and leads to unusual intensification of pain that is out of proportion to the inciting stimulus. For example, light touch from clothing on the skin is perceived as intensely painful. Central sensitization is also thought to contribute to the spreading of pain to other body sites in several chronic pain disorders.

In chronic pain disorders, the function of the central descending inhibitory modulating system is likely impaired and is traditionally measured by a phenomenon identified as "conditioned pain modulation (CPM)" and more recently measured by a phenomenon of "offset analgesia" (OA). The OA test is more robust than the CPM test and likely more acceptable to most patients, especially children, because it is shorter in duration and uses a more tolerable painful stimulus. Compared to CPM, the OA test is more tolerable because it is conducted using a painful test stimulus that is less than the maximal (suprathreshold). Additionally, the time of exposure to the painful stimulus is significantly shorter, a few seconds, in the OA test compared to CPM.

The central descending inhibitory pathway that modulates pain as tested by OA is functional and mature in healthy children as young as 6 year of age, but it has yet to be investigated in children with chronic pain disorders. The investigators plan to test OA responses in a population of common pediatric pain disorders with overlapping symptomology attributed to central sensitization (such as chronic musculoskeletal pain, chronic abdominal pain and chronic headaches and chronic regional pain syndromes) and compare their responses with an age- and sex-matched control group. The characteristics of OA responses in each group will allow for assessment of the presence or absence of central sensitization as a mechanism driving the persistent, abnormal pain in a subgroup of these chronic pain disorders. The investigators hypothesize that central sensitization is the potential contributory mechanism of the central nervous system heightened sensitivity to two testing stimuli of painful (moderate heat discomfort sensation) and non-painful (warmth sensation) in children with chronic pain disorders. These types of sensations mimic those that children would be expected to experience their natural environment during typical activities of daily living such as showering/bathing in warm water or hand washing.

Additionally, the Pain Sensitivity Questionnaire (PSQ) and Central Sensitization Inventory (CSI) will be used as clinical screening tools for subjective report of sensitization symptoms, and are simple and easy to administer in a clinical setting. The investigators hypothesize that these measures will correlate with the objective offset analgesia responses thus allowing for assessment of central sensitization in children with chronic pain disorders.

These tests are advantageous because they are feasible to perform rapidly in a clinic setting and have utility for measurement of patient responses to therapeutic interventions. If this concept is supported by this study, future studies could utilize OA to examine the effects of various pharmacological and physical interventions used to manage children with chronic pain disorders including intensive interdisciplinary rehabilitation or specific interventions such as aerobic exercise, which likely modulates pain via similar mechanisms.

DETAILED DESCRIPTION:
Specific Aims/Objectives To date, OA has not been evaluated in pediatric chronic pain disorders. In the current study, the investigators plan to measure OA responses in a population of common pediatric pain disorders. The primary objective of this study is to determine if OA paradigm can detect impairment of central inhibitory modulation pathways in subgroups of chronic pain disorders in children and adolescents. The investigators hypothesize that chronic pain in children and adolescents results from central sensitization and impaired central inhibitory modulation of pain and thus children with chronic pain disorders will have a decreased OA response compared with healthy controls. If the results of this study are positive, this testing paradigm could be a valuable objective marker in examining the efficacy of pharmacological and/or rehabilitative treatment modalities in reversing or alleviating central sensitization-induced pain in children with chronic pain disorders. Additionally, if existing self-report questionnaires, Pain Sensitivity Questionnaire (PSQ) and Central Sensitivity Inventory, correlate with the magnitude of offset analgesia observed, they could be used to screen for central sensitization in high volume and busy clinical settings.

Aim 1: To determine if children with common chronic pain disorders, including musculoskeletal pain, complex regional pain syndrome, functional abdominal pain and chronic headaches demonstrate impaired ability to actuate central descending inhibitory function as measured by a test of offset analgesia.

To accomplish this aim, the investigators will compare 30 children with common chronic pain disorders with 30 age and sex matched controls. Power will be 80% to detect a 20% or larger difference in the change in self-reported pain scores as a result of the dynamic heat pain test stimulus between the two groups using a Student t-test (nQuery Advisor version 7.0, Statistical Solutions, Cork, Ireland).

Aim 2: To determine if the Pain Sensitivity Questionnaire (PSQ) and/or Central Sensitization Inventory (CSI) can serve as screening tools for assessment of central sensitization i.e., impairment of central descending inhibitory function in children with common chronic pain disorders.

To accomplish this aim investigators will correlate scores on the above scales with the magnitude of offset analgesia using Pearson correlations in 30 children with chronic pain disorders and 30 healthy age and sex-matched controls. The investigators hypothesize that the magnitude of OA will correlate with either PSQ, CSI or both thus these questionnaires would serve as assessment tools for central sensitization in children with common chronic pain disorders in clinical setting. The Mann-Whitney U-test will be applied to compare medians and interquartile ranges on the PSQ and CSI between the chronic pain and healthy control groups. In addition, investigators will identify individuals who show a decrease in VAS pain scores after the dynamic test stimulus of at least 20% (responders) and will assess whether PSQ and CSI can predict responders and non-responders using a receiver operating characteristic (ROC) curve approach with area under the curve (AUC) to measure how well pain perception and central sensitization assessment tools can help to identify responders and non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing chronic pain defined as pain persisting for 3 months.
* Ages 10-17 years, both sexes and all races and ethnic groups.
* Patients with moderate pain rated as 5/10 and greater on a numeric rating scale of 0 to 10 points.
* English speaking.
* If patients are taking medications such as psychotropic (e.g., SSRI), opioid, anxiolytics or anticonvulsive drugs for pain such as gabapentinoids, they must be on stable doses for at least one week.
* Stable anxiety and depression.

Exclusion Criteria:

* Intermittent pain or pain of less than 3-month duration.
* Allodynia in the upper extremities
* Patients with poor understanding of English language or developmental disorders that affect the ability to reliably rate pain, read questionnaires and follow study instructions.
* Children and adolescents with a history of central nervous system, heart, kidney, liver, and respiratory system diseases.
* Psychiatric disorders such as conversion, bipolar disorder or psychosis.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Response to Offset analgesia stimulus | outcome will be observed in a single session over one hour period
  A reduction in self-reported pain intensity when a moderate heat-pain stimulus is applied for 5 seconds, raised by 1 degree C for 5 seconds, reduced by 1 degree C, and held for 20 seconds. During all tests, patients will rate heat pain intensity continuously in real time using the linear, electronic visual analogue scale (eVAS). Patients will use their dominant hand to operate sliding knob of the eVAS with the following two anchors on 0 to 100 mm line. The left endpoint designated as "no pain sensation" (0 mm) and the right endpoint as "most intense pain sensation imaginable" (100 mm).

SECONDARY OUTCOMES:
Response to a Controlled Stimulus | outcome will be observed in a single session over one hour period
  A reduction in self-reported pain intensity when a moderate heat-pain stimulus is applied for 5 seconds, raised by 1 degree C for 5 second, reduced to 32 degree C, and held for 20 seconds. During all tests, patients will rate heat pain intensity continuously in real time using the linear, electronic visual analogue scale (eVAS). Patients will use their dominant hand to operate sliding knob of the eVAS with the following two anchors on 0 to 100 mm line. The left endpoint designated as "no pain sensation" (0 mm) and the right endpoint as "most intense pain sensation imaginable" (100 mm).
Response to a Constant Stimulus | outcome will be observed in a single session over one hour period
  A reduction in self-reported pain intensity when a moderate heat-pain stimulus (test temperature) is applied 30 seconds. During all tests, patients will rate heat pain intensity continuously in real time using the linear, electronic visual analogue scale (eVAS). Patients will use their dominant hand to operate sliding knob of the eVAS with the following two anchors on 0 to 100 mm line. The left endpoint designated as "no pain sensation" (0 mm) and the right endpoint as "most intense pain sensation imaginable" (100 mm).
Pain sensitivity questionnaire | outcome will be observed in a single session over one hour period
  Self reported pain intensity of imagined painful events in their daily activities. Participants are instructed to rate how painful each situation would be for them on a numeric rating scale ranging from 0 ( = not painful at all) to 10 ( = worst pain imaginable). The total score is derived as an average of sum of each response with higher scores indicating higher pain sensitivity.
Central sensitization inventory | outcome will be observed in a single session over one hour period
  Self reported instrument for screening possible presence of central sensitization. Responses are recorded for the frequency of each symptom on a Likert scale from 0 (never) to 4 (always), resulting in a total possible score of 100. Higher scores are associated with a higher degree of self-reported symptomology.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No